CLINICAL TRIAL: NCT04095715
Title: Diagnosis of Platelet Dense Granules Anomalies in Unexplained Hemorrhagic Syndromes
Brief Title: Anomalies of Dense Platelet Granules
Acronym: AGRAD
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Assistance Publique Hopitaux De Marseille (Other); CENTRE DE REFERENCE DES MALADIES HEMORRAGIQUES CONSTITUTIONNELLES (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP190393
Record Dates: First submitted 2019-06-18; First posted 2019-09-19 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Spontaneous Induced Unexplained Haemorrhagic
Keywords: Dense platelet granules; Thrombopathy; Hemorrhagic symptomatology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children and adults with unexplained hemorrhagic syndrome: Patients with spontaneous or induced hemorrhagic manifestations who are present for a consultation to investigate a thrombopathy or during follow-up consultations as part of their usual care.
  Interventions: Other: Haemostasis consultation; Biological: Standard management of patients suspected of thrombopathy

INTERVENTIONS:
Other: Haemostasis consultation — Haemostasis consultation
Biological: Standard management of patients suspected of thrombopathy — Standard management of patients suspected of thrombopathy

SUMMARY:
The study aims to know the overall prevalence of granular deficits and their breakdown by type (anomaly of number, content or secretion) in a population of patients with hemorrhagic symptomatology after exclusion of other known causes.

This study consists also to evaluate the association between the presence of a deficit in dense granules and (1) the intensity of the hemorrhagic phenotype (hemorrhagic score) (2) the nature of hemorrhages (post-operative, spontaneous, atypical...)

-Evaluate the association between the type of deficit in dense granules and (1) the intensity of the hemorrhagic phenotype (hemorrhagic score) (2) the nature of hemorrhages (post-operative, spontaneous, atypical...)

DETAILED DESCRIPTION:
Patients will be recruited during the exploration visit (v0) or the confirmation/typing visit (v1) according to their follow-up.

* Exploration visit (v0): inclusion of patients without prior platelet exploration, and study of their dense platelet granules.
* Confirmation/typing visit (v1): verification of the persistence of anomalies detected in patients with an abnormality identified during v0 (no later than 6 months after v0) and in patients for whom a dense granules anomaly has already been identified during their standard management prior to the start of the study. Completion of complementary examinations to complement the typing of the granular anomaly and molecular analysis for family cases

ELIGIBILITY:
Inclusion Criteria:

* Adult or child patient ≥ 2 years
* Having a hemorrhagic score ISTH > 3 for men, > 5 for women and > 2 for children.
* With no abnormal coagulation (defined by normal TP and TCK or activity ≥ 50% of FII, FV, FVII, FX, FVIII, FIX, FXI)
* no deficiency of Willebrand factor (defined by a cofactor activity with Ristoctin (VWF: RCo < 50%))
* no a known major thrombocytopenia/thrombopathy linked to a deficiency of one of the major platelet receptors
* Information of the patient and/or his legal representative present

Exclusion Criteria:

* Inability or refusal of compliance with research requirements
* Thrombocytopenia < 100 G/L
* Treatments interfering with platelet functions within 10 days prior to inclusion
* Malignant hemopathy

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients addressed to the specialized haemostasis consultations of the various services associated with the project for the exploration of haemorrhagic symptomatology referring to a primary haemostasis anomaly.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Platelet response to different agonists | Baseline (M0)
  Us of some low-dose agonists such as ADP, epinephrine or collagen, which are particularly susceptible to granular defects, on platelet-rich plasma (PRP) prepared from the patient's blood sample to be explored
Platelet response to different agonists | At 6 months
  Use of some low-dose agonists such as ADP, epinephrine or collagen, which are particularly susceptible to granular defects, on platelet-rich plasma (PRP) prepared from the patient's blood sample to be explored
Granular Delta content | Baseline (M0)
  Dosage of platelet serotonin by measuring platelet serotonin by HPLC.
Measurement of ATP | Baseline (M0)
  The measurement is based on the principle of bioluminescence with a two-step transformation reaction of luciferin in the presence of luciferase, this reaction requiring the presence of ATP
Measurement of ATP | At 6 months
  The measurement is based on the principle of bioluminescence with a two-step transformation reaction of luciferin in the presence of luciferase, this reaction requiring the presence of ATP
Measurement of granules opacity | Baseline (M0)
  Delta granules contain calcium, which makes them naturally opaque to electrons and thus allows their direct visualization in electronic microscopy.
Measurement of granules opacity | at 6 months
  Delta granules contain calcium, which makes them naturally opaque to electrons and thus allows their direct visualization in electronic microscopy.

SECONDARY OUTCOMES:
Hemorrhagic risk assessment | Baseline (M0)
  Evaluation using the ISTH score
Typage of delta granules anomalies | At 6 months
  Fib-SEM technic by focussed ion beam scanning which allows a 3D reconstitution of the platelets and thus to visualize any empty granules
Genetic anomalies of delta granules | At 6 months
  Sequencing on a broad set of genes involved in platelet function. Bioinformatic analysis is carried out using BWA-MEM software (Alignment on the genome version HG19)
Prothrombin consumption | Baseline (M0)
  Evaluated by% of residual Thrombin after plasma coagulation
Prothrombin consumption | at 6 months
  Evaluated by% of residual Thrombin after plasma coagulation

CONTACTS AND LOCATIONS:
Overall Officials: Delphine BORGEL, PhD, Principal Investigator — APHP
Locations (1):
- Hôpital Necker Enfants Malades - AP-HP, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gresele P, Harrison P, Bury L, Falcinelli E, Gachet C, Hayward CP, Kenny D, Mezzano D, Mumford AD, Nugent D, Nurden AT, Orsini S, Cattaneo M. Diagnosis of suspected inherited platelet function disorders: results of a worldwide survey. J Thromb Haemost. 2014 Sep;12(9):1562-9. doi: 10.1111/jth.12650. Epub 2014 Jul 25. PMID 24976115
- [Background] Quiroga T, Goycoolea M, Panes O, Aranda E, Martinez C, Belmont S, Munoz B, Zuniga P, Pereira J, Mezzano D. High prevalence of bleeders of unknown cause among patients with inherited mucocutaneous bleeding. A prospective study of 280 patients and 299 controls. Haematologica. 2007 Mar;92(3):357-65. doi: 10.3324/haematol.10816. PMID 17339185
- [Background] Fiore M, Garcia C, Sié P, et al. δ-storage pool disease: an underestimated cause of unexplained bleeding. Hématologie 2017-8; 243-254.
- [Background] Gresele P; Subcommittee on Platelet Physiology of the International Society on Thrombosis and Hemostasis. Diagnosis of inherited platelet function disorders: guidance from the SSC of the ISTH. J Thromb Haemost. 2015 Feb;13(2):314-22. doi: 10.1111/jth.12792. Epub 2015 Jan 22. No abstract available. PMID 25403439
- [Background] Mumford AD, Frelinger AL 3rd, Gachet C, Gresele P, Noris P, Harrison P, Mezzano D. A review of platelet secretion assays for the diagnosis of inherited platelet secretion disorders. Thromb Haemost. 2015 Jul;114(1):14-25. doi: 10.1160/TH14-11-0999. Epub 2015 Apr 16. PMID 25879272
- [Background] Selle F, James C, Tuffigo M, Pillois X, Viallard JF, Alessi MC, Fiore M. Clinical and Laboratory Findings in Patients with delta-Storage Pool Disease: A Case Series. Semin Thromb Hemost. 2017 Feb;43(1):48-58. doi: 10.1055/s-0036-1584568. Epub 2016 Jun 15. PMID 27304079